CLINICAL TRIAL: NCT03247712
Title: Neoadjuvant Immunoradiotherapy: Head & Neck Cancer (NIRT-HNC)
Brief Title: Neoadjuvant Immunoradiotherapy in Head & Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIRT-HNC
Record Dates: First submitted 2017-08-08; First posted 2017-08-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; radiation; surgery; phase 1; immunotherapy; nivolumab; antibodies
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment Cohort 1 (Experimental): Nivolumab administration (3 doses) and radiation (5 days) therapy prior to restaging and surgical resection followed by additional administration of nivolumab (3 doses).
  Interventions: Drug: Nivolumab; Procedure: Surgical Resection; Radiation: Radiation (5 days)
- Treatment Cohort 2 (Experimental): Nivolumab administration (3 doses) and radiation (3 days) therapy prior to restaging and surgical resection followed by additional administration of nivolumab (3 doses).
  Interventions: Drug: Nivolumab; Procedure: Surgical Resection; Radiation: Radiation (3 days)
- Treatment Cohort 3 (Experimental): Radiation (3 days) therapy prior to restaging and surgical resection followed by additional administration of nivolumab (3 doses).
  Interventions: Drug: Nivolumab; Procedure: Surgical Resection; Radiation: Radiation (3 days)
- Treatment Cohort 4 (Experimental): Nivolumab administration (3 doses) and radiation (3 days) therapy prior to restaging and surgical resection followed by additional administration of nivolumab (3 doses).
  Interventions: Drug: Nivolumab; Procedure: Surgical Resection; Radiation: Radiation (3 days)

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240mg IV q2wks or 480mg IV q4wks
  Other Names: Opdivo
Procedure: Surgical Resection — Surgical Resection of Tumor
Radiation: Radiation (5 days) — 8Gy x 5 (Mon-Fri) GTV+3mm
  Arms: Treatment Cohort 1
Radiation: Radiation (3 days) — 8Gy x 3 (Monday, Wednesday, Friday) GTV+3mm
  Arms: Treatment Cohort 2; Treatment Cohort 3; Treatment Cohort 4

SUMMARY:
The purpose of this study is to test the safety of neoadjuvant immunoradiotherapy as a safe means of down-staging Head and Neck Squamous Cell Carcinoma (HNSCC) prior to surgical resection.

DETAILED DESCRIPTION:
This clinical trial uses nivolumab and radiotherapy prior to definitive surgical resection of tumors in patients with Head and Neck Squamous Cell Carcinoma (OHNSCC) with the primary objective of determining the safety and feasibility of preoperative immunoradiotherapy. In addition, tumor tissue, microbiome samples, and peripheral blood will be obtained for exploratory immunologic end points including measurements of tumor infiltrating immune cell populations based on flow cytometry and immunohistochemistry as well as circulating immunological parameters. This is the first study to evaluate the safety and efficacy of neoadjuvant radiation + PD-1 blockade in patients with HNSCC.

Estimated duration of 20 weeks: neoadjuvant immunoradiotherapy +/- surgery, followed by 6 doses of nivolumab 480mg IV q4wks +/- risk-adapted adjuvant therapy, per standard of care.

Phase I safety lead-in study (n = 6) evaluating the safety of neoadjuvant immunoradiotherapy in HNSCC, followed by phase II efficacy study (n = 28, total) to assess rate of down-staging after neoadjuvant immunoradiotherapy using Simon's two-stage design (futility assessment at n = 12).

The phase 1 portion of this study will require 6 patients and is therefore expected to complete in 6 months. Although non-surgical patients are eligible to enroll, they will not be counted toward accrual for either the primary safety endpoint, (as by definition, unplanned delay of surgery cannot exist); nor the secondary efficacy endpoint, as potential for surgical staging is absent.

So long as 2 or fewer surgical delays are observed (primary safety endpoint), the phase 2 portion of study will proceed (secondary efficacy endpoint). Patients will be followed for disease free and overall survival at 5 years.

Eligible patients may be enrolled unless a rate of unplanned surgical delay attributed to immunoradiotherapy is found to exceed 33% after enrollment of the first 6 patients. We estimate 10 to 20 patients per year will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with squamous cell carcinoma of the head and neck region, (including mucosal,cutaneous, or nodal) who are planned for surgical resection and in the opinion of the investigator are able to safely undergo neoadjuvant anti-PD-1 and radiation. In addition, the following are eligible (but will not contribute toward total accrual): non-surgical cases that are planned for palliative RT or that refuse or are unfit for definitive concurrent chemotherapy.
2. HPV status as determined by p16 immunostain
3. Cohort 3: HPV-positive patients only
4. Cohort 4: HPV-negative patients only
5. Age 18 years or above with ability to give informed consent, comply with the protocol, and sign a study-specific consent document. Patients with history of psychiatric illness must be judged by the investigator as able to understand the investigational nature and risks associated with the therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status deemed suitable by investigator for study requirements.
7. Laboratory values (most recent), must be within 6 weeks of week 0 on study:

   * WBC ≥ 2000/uL, ANC ≥ 1000/uL
   * Hgb > 8g/dL (patients may be transfused to reach this level)
   * Platelets > 50,000 cells/mm3
   * Creatinine ≤ 3 x ULN
   * AST/ALT ≤ 5 x ULN for subjects without liver metastasis; or ≤ 8 x ULN for subjects with liver metastasis, [per investigator brochure]
   * Total bilirubin ≤ 3 x ULN, (except subjects with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
   * Negative pregnancy test (bHCG urine or serum, women of childbearing potential only)
8. Women of child-bearing potential (WOCBP) must agree to follow adequate contraceptive practices to avoid pregnancy for the duration of treatment with nivolumab plus 5 half-lives of nivolumab (75 days) plus 30 days (duration of ovulatory cycle) for a total of 105 days post-treatment completion.
9. Males who are sexually active with WOCBP must agree to follow adequate contraceptive practices to avoid pregnancy for the duration of treatment with study drug (s) plus 5 half lives of the study drug (75 days) plus 90 days (duration of sperm turnover) for a total of 165 days post-treatment completion.

Exclusion Criteria:

1. Any clinical factors such as bleeding, active infection, or psychiatric factors that in the judgment of the investigator would preclude safe participation and compliance with study procedures.
2. HNSCC for which radiation is not indicated during normal treatment course.
3. Need for chronic maintenance with oral steroids ≥20mg daily prednisone equivalent; inhaled, topical or non-absorbed steroids are acceptable.
4. History of or current active autoimmune disease, [e.g. including but not limited to inflammatory bowel diseases [IBD], rheumatoid arthritis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barre syndrome)], which in the judgment of the investigator poses an active and significant morbidity risk. Vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism are not exclusionary. Patient and investigator may opt to accept risk of autoimmune disease flare, based on shared-decision making with consideration of risk/benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an Unplanned Delay to Surgery [Safety and Tolerability of Neoadjuvant Treatment] | 6 weeks
  Safety endpoint: Number of patients with an Unplanned Delay to Surgery defined as any change to scheduled surgery date considered to be at least possibly related to neoadjuvant treatment.

SECONDARY OUTCOMES:
Number of patients with decrease in tumor size or number of lymph nodes involved [Efficacy of Neoadjuvant Treatment] | 6 weeks
  Efficacy endpoint: Number of patients with decrease in tumor size of greater than 10% or decrease in the number of lymph nodes involved by 10% by week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Rom Leidner, MD, Principal Investigator — Providence Health and Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leidner R, Crittenden M, Young K, Xiao H, Wu Y, Couey MA, Patel AA, Cheng AC, Watters AL, Bifulco C, Morris G, Rushforth L, Nemeth S, Urba WJ, Gough M, Bell RB. Neoadjuvant immunoradiotherapy results in high rate of complete pathological response and clinical to pathological downstaging in locally advanced head and neck squamous cell carcinoma. J Immunother Cancer. 2021 May;9(5):e002485. doi: 10.1136/jitc-2021-002485. PMID 33963014
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/